CLINICAL TRIAL: NCT03575325
Title: A Single-Arm, Open-Label Phase 2 Pilot Study of Vyxeos (CPX-351) in Adults With Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: Vyxeos(CPX-351) in Adults w R/R Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19482
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Lymphoid Leukemia; Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia; Relapsed Acute Lymphoblastic Leukemia
Keywords: T-cell acute lymphoblastic leukemia; B-cell acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia, Lymphoid; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — CPX-351

STUDY DESIGN:
Intervention Model Description: This is an open label, single arm, single center, phase 2 pilot study of Vyxeos induction & consolidation in relapsed and refractory ALL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CPX-351 Treatment (Experimental): Participants will receive induction with CPX-351 at a dose of 100 u/m^2 administered intravenously over 90 minutes on days 1, 3 and 5 of a 28 day cycle.
  This may be followed by consolidation with CPX-351 at a dose of 65 u/m^2 administered intravenously over 90 minutes on days 1 and 3 of a 28 day cycle (up to 3 cycles).
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351 — The infusion of CPX-351 (cytarabine:daunorubicin) Liposome Injection will be performed through a central venous catheter, using an infusion pump to ensure that the drug is infused over the specified time period.
  Other Names: Vyxeos; cytarabine:daunorubicin

SUMMARY:
This study involves Vyxeos (CPX-351), a formulation of a fixed combination of the two anti-tumor drugs, cytarabine and daunorubicin that will be given as an infusion over 90 minutes. This study will use what is called a "liposome" injection. This is a special fat capsule (called a liposome) that surrounds the cytarabine and daunorubicin and protects the drugs from being eliminated/destroyed by the body.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent/assent for the trial.
* Be ≥ 18 years of age on day of signing informed consent.
* Able to adhere to the study visit schedule and other protocol requirements.
* Pathologically confirmed B- or T-cell acute lymphoblastic or mixed phenotype acute leukemia, with >5% peripheral blood or bone marrow lymphoblasts and/or extramedullary disease >1x1cm.
* Relapsed or refractory acute lymphoblastic leukemia after at least 1 prior cycle of therapy. Patients with Philadelphia chromosome positive disease must have failed at least two prior tyrosine kinase inhibitors.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Cardiac ejection fraction ≥ 50% by echocardiography or multigated acquisition scan (MUGA).
* Must be at least 2 weeks out from any prior systemic chemotherapy, blinatumumab, radiation, and/or other investigational agents, and have recovered to grade 1 from any toxicity related to prior therapy. Glucocorticoids are permitted up to 1 day prior to the first dose.
* Serum bilirubin and creatinine less than 1.5x upper limit of normal (ULN). AST and ALT must be less than 3x ULN, unless there is suspected liver involvement.
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test at screening. A FCBP is considered when a sexually mature female: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months.
* A FCBP must agree to use of two methods of highly effective contraception, be surgically sterile, or abstain from heterosexual activity for the course of the study through 30 days after the last dose of study treatment.
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 30 days after the last dose of study therapy. Men must agree to not donate sperm during and after the study

Exclusion Criteria:

* Clinical evidence of active central nervous system (CNS) leukemia.
* Any major surgery or radiation therapy within four weeks.
* Any active infection requiring systemic therapy, including HIV, Hepatitis B, and/or Hepatitis C.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator (including but not limited to severe graft-versus-host disease, unstable angina, pulmonary hypertension, active/prior veno-occlusive disease of the liver or severe CHF (NYHA III-IV).
* Patients with active (uncontrolled, metastatic) second malignancies.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 30 after the last dose of trial treatment.
* Hypersensitivity to cytarabine, daunorubicin, or liposomal products.
* History of Wilson's disease or other copper-metabolism disorder.
* Patients with prior cumulative anthracycline exposure of greater than 368 mg/m^2 daunorubicin or equivalent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bijal Shah, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CPX-351 Treatment: Participants will receive induction with CPX-351 at a dose of 100 u/m^2 administered intravenously over 90 minutes on days 1, 3 and 5 of a 28 day cycle.
  This may be followed by consolidation with CPX-351 at a dose of 65 u/m^2 administered intravenously over 90 minutes on days 1 and 3 of a 28 day cycle (up to 3 cycles).
  CPX-351: The infusion of CPX-351 (cytarabine:daunorubicin) Liposome Injection will be performed through a central venous catheter, using an infusion pump to ensure that the drug is infused over the specified time period.
Period: Overall Study
Arm/Group | CPX-351 Treatment
Started | 11
Completed | 10
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | CPX-351 Treatment
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate (CR) + CR With Incomplete Recovery (CRi)
Description: Expansion from phase II pilot to a phase II trial will depend on demonstration of CR/CRi amongst 4 of the initial 10 treated patients. Investigators will measure remission rate at day 28 to address the primary endpoint of complete remission (with or without complete hematologic recovery), as defined by Cheson Criteria (ref 27). For those with extramedullary disease, Lugano criteria will be used to assess response. This is a standard assessment of drug efficacy for phase 2 clinical trial design in acute leukemias, as response correlates closely with progression free- and overall survival (PFS and OS).
Time Frame: At day 28
Population: Evaluable participants
Measure: Number; unit: Percent of participants
Arm/Group | CPX-351 Treatment
Number analyzed (Participants) | 10
Percent of participants | 30

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival as defined by Cheson and Lugano Criteria, namely progression, failure to respond, or death, as assessed from time of first treatment. Progression Free Survival will be reported as per Cheson Criteria, and analyzed using a standard Kaplan-Meier approach. Patients will undergo bone marrow biopsy evaluation after each cycle of therapy per standard of care to facilitated assessment.
Time Frame: 12 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CPX-351 Treatment
Number analyzed (Participants) | 10
Days | 57 [10 to 105]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival as defined by Cheson and Lygano Criteria, namely death due to any cause as assessed from time of first treatment. Overall Survival will be reported as per Cheson Criteria, and analyzed using a standard Kaplan-Meier approach. Patients will undergo bone marrow biopsy evaluation after each cycle of therapy per standard of care to facilitated assessment.
Time Frame: 12 months
Population: Evaluable participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | CPX-351 Treatment
Number analyzed (Participants) | 10
Days | 218 [161 to 275]

4. Secondary Outcome: Minimal Residual Disease (MRD)
Description: MRD assessment will be provided using ClonoSeq test result. ClonoSEQ® is an FDA-cleared test used to detect minimal residual disease (MRD) in bone marrow from patients with multiple myeloma or B-cell acute lymphoblastic leukemia (B-ALL) and blood or bone marrow from patients with chronic lymphocytic leukemia (CLL).
Time Frame: At day 28
Population: Evaluable participants - Participants who achieved CR or CRi
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351 Treatment
Number analyzed (Participants) | 3
Participants
  No trackable clone by ClonoSeq | 2
  Complete Molecular Remission by ClonoSeq | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent until 30 days after the last dose of CPX-351, approximately 34 months.
Groups:
- CPX-351 Treatment Induction Dose: Participants who received induction with CPX-351 at a dose of 100 u/m^2 administered intravenously over 90 minutes on days 1, 3 and 5 of a 28 day cycle.
- CPX-351 Treatment Induction Dose + 1 Consolidation Dose: Participants who received induction with CPX-351 at a dose of 100 u/m^2 administered intravenously over 90 minutes on days 1, 3 and 5 of a 28 day cycle. Participants then received one consolidation dose of CPX-351 at a dose of 65 u/m^2 administered intravenously over 90 minutes on days 1 and 3 of a 28 day cycle
- CPX-351 Treatment +2 Consolidation Doses: Participants who received induction with CPX-351 at a dose of 100 u/m^2 administered intravenously over 90 minutes on days 1, 3 and 5 of a 28 day cycle. Participants then received two consolidation doses of CPX-351 at a dose of 65 u/m^2 administered intravenously over 90 minutes on days 1 and 3 of a 28 day cycle
Arm/Group | CPX-351 Treatment Induction Dose | CPX-351 Treatment Induction Dose + 1 Consolidation Dose | CPX-351 Treatment +2 Consolidation Doses
All-Cause Mortality (participants affected / at risk) | 1/7 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPX-351 Treatment Induction Dose (N=7) | CPX-351 Treatment Induction Dose + 1 Consolidation Dose (N=3) | CPX-351 Treatment +2 Consolidation Doses (N=1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Cellulitis of right foot
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPX-351 Treatment Induction Dose (N=7) | CPX-351 Treatment Induction Dose + 1 Consolidation Dose (N=3) | CPX-351 Treatment +2 Consolidation Doses (N=1)
Abdominal Pain (Gastrointestinal disorders) | 4 (7) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (6) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (3) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (19) | 2 (16) | 1 (6)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (7) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — hypovolemia
Blood bilirubin increased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) — Myopericarditis
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 3 (5) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (2) | 2 (3) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders -Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — subconjuctival hemorrhage, right
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6) | 2 (2) | 1 (2)
Fever (General disorders) | 1 (7) | 2 (2) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 1 (3) | 2 (6) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (8) | 3 (6) | 1 (1)
Hematoma (Vascular disorders) | 2 (3) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (5) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (8) | 1 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Immune system disorders - other (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — hypogammaglobulinemia
Infections and infestations - Other (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (2) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (3) | 0 (0) | 0 (0)
Investigations - Other (Investigations) | 1 (1) | 1 (3) | 0 (0)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (2)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (5) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 3 (7) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (17) | 3 (16) | 1 (7)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Pain (General disorders) | 1 (2) | 3 (8) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 6 (24) | 3 (31) | 1 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (7) | 2 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders -Other (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Serum amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Skin infection (Infections and infestations) | 2 (5) | 0 (0) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cardiac troponin T increased (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — soft tissue mass
Nervous system disorders - Other (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) — Subarachnoid hemorrhage
GGT Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT03575325/Prot_SAP_000.pdf